CLINICAL TRIAL: NCT02993692
Title: Nasotracheal Intubation in Children for Outpatient Dental Surgery: Is Fiberoptic Bronchoscopy Useful?
Brief Title: Nasotracheal Intubation in Children for Outpatient Dental Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, M.D., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Asozkan
Record Dates: First submitted 2016-12-01; First posted 2016-12-15 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Nasotracheal Intubation
Keywords: direct laryngoscopy; fiberopitc bronchoscopy; nasotracheal intubation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fiberoptic bronchoscopy (Other): I want to see the difference between the two group about hemodynamic and intraoculer pressure responses about fiberoptic bronchoscopy.
  Interventions: Device: Direct laryngoscopy and fiberoptic bronchoscopy
- direct laryngoscopy (Other): I want to see the difference between the two group about hemodynamic and intraoculer pressure responses about direct laryngoscopy.
  Interventions: Device: Direct laryngoscopy and fiberoptic bronchoscopy

INTERVENTIONS:
Device: Direct laryngoscopy and fiberoptic bronchoscopy — These devices is used in endotracheal intubation and tonopen for measuring of intraoculer pressure. I want to see whcih is better.
  Other Names: tonopen

SUMMARY:
The aim of study was to compare the hemodynamic responses and adverse events associated with nasotracheal intubation (NTI) using a fiberoptic bronchoscope (FOB) and a direct laryngoscope (DLS) in children undergoing general anesthesia for outpatient dental surgery. Eighty children (aged 5-15 years) were scheduled to undergo outpatient dental surgery under general anesthesia and who required nasotracheal intubation were included.

DETAILED DESCRIPTION:
Investigators obtained confirmation from the Inonu University Medical Faculty Hospital Ethics Committee (2015/101) and written informed consent from the guardians of all 80 children. These children, who had a American Society of Anesthesia physical status of I-II, had a Mallampati Score of 1-2, were aged 5-15 years, were scheduled to undergo outpatient dental surgery under general anesthesia, and required nasotracheal intubation were included in this prospective and randomized study. Exclusion criteria included the following: the patient's refusal for study consent, active upper respiratory infection, airway abnormalities, nasal mass or nasal injury, bleeding disorders, allergies to anesthetics, uncontrolled hypertension, morbid obesity, hepatic or renal failure, cardiovascular diseases, a history of nasopharyngeal surgery and those who were difficult to intubate. Children were randomly assigned into the direct laryngoscopy group (n = 40) or the fiberoptic bornchoscopy group (n = 40) according to a computer-randomized table. General anesthesia was administered to children due to the learning difficulties. The number of models was decided by a statistical power analysis after the conclusions from the pretest were obtained. All children fasted at least for 6 h before surgery, and the oral intake of clear fluids was restricted for 2-3 h. Premedication of midazolam (0.5 mg/kg) was orally administered in apple juice (0.5 mL/kg of body weight) 1 h prior to anesthesia. After being admitted to the operating room, the patient's systolic blood pressure (SBP) and heart rate (HR) were continually monitored with a multichannel physiologic monitor and the baseline values for SBP and HR were recorded. Thirty min before the intubation attempt, the nasal mucosa of both nostrils were anesthetized with a topical vasoconstrictor (0.05% xylometazoline spray, and 2% lidocaine 1 mL two times in each nostril) (9) to attenuate cardiovascular responses and adverse events in all children. Anesthesia was induced with 8% sevoflurane with eight deep breaths via a face mask, and the patient was maintained on 4% end-tidal sevoflurane, fentanyl 2 µr/kg and rocuronium 0.6 mg/kg. NTI was achieved 2 min after rocuronium injection. The more patent nostril was selected for intubation. An experienced anesthetist performed all intubations in the study and an assistant applied the maneuvers (jaw trust) and evaluated the patient during the postoperative visits. All NTIs, both DLS and FOB, were conducted by the same experienced anesthetist (the anesthetist had performed DLS and the FOB nasal intubation in more than 150 patients, including in at least 100 children before the study). A study nurse documented the anesthetic data and timing. In the DLS group, the spiral tube was inserted into the nose and intubated with a Macintosh laryngoscope according to conventional procedures using Magill forceps. In the FOB group, NTI was conducted using an FOB with an outer diameter of 3.1 mm through the selected clear nasal passage with a spiral tracheal tube. The appropriate size of the tracheal tube for a child was determined with the following formula (10): Internal diameter (mm) = age/3 + 3.5 in both groups. The same type of tube was used in each group. Before intubation, enough lidocaine gel was placed on the tracheal tube, and the FOB was guided into patients with a suitable spiral tracheal tube. All tracheal tubes were cuffed and heat-softened in warm normal saline and lubricated to reduce mechanic stimuli to airway structures. During the intubation, the head of the patient was the in supine position, and an assistant applied a jaw thrust for opening the nasopharyngeal passage and improved the image in all patients in the FOB group. If indicated (a suboptimal laryngeal view or resistance in passing of the tracheal tube), anterior laryngeal pressure and tongue withdrawal by digital traction was performed to improve the laryngeal field of view. When the glottis was clearly visible, the FOB was advanced through the vocal cords, and jaw thrust movement was released. To prevent the stimulation of the carina, the tube was placed 4 cm below the glottis, sliding over the FOB. Intubation was verified with the FOB, and end-tidal CO2 concentrations at 35-40 mmHg were monitored. A throat pack was inserted by the anesthetist after the measurements were taken. Anesthesia was maintained with 2% sevoflurane and 50% N20 in oxygen with 1.5 l min-1 fresh gas flow and 35-40 mmHg end-tidal CO2 concentrations. Isolyte-P was administered at rate of 15 mL/kg/h IV, and acetaminophen (15 mg kg-1) was infused for postoperative analgesia in all children.

SBP and HR were recorded at baseline, after induction of anesthesia, at the time of intubation, and 1, 3 and 5 min after intubation. The intubation time (the time from when manual ventilation with a facemask stopped to restarting ventilation via the nasotracheal tube and when carbon dioxide (CO2) was detected by capnography) was recorded by another anesthetist with a digital stopwatch. Nose bleeding after intubation (epistaxis), laryngospasms, bradycardia (HR<65 beat min-1), hypoxic episodes (SpO2<90%) and the surgery type were also recorded. Adverse events (hoarseness, sore throat) were assessed 24 h after surgery. If a sore throat developed, additional analgesics were not administered. If bradycardia or desaturation (SpO2<90%) occurred for more than 2 min, the intubation was interrupted, and patients were ventilated with 100% oxygen and were administered IV atropine (5-10 µg / kg).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status of I-II, had a Mallampati Score of 1-2, were aged 5-15 years, were scheduled to undergo outpatient dental surgery under general anesthesia

Exclusion Criteria:

* The patient's refusal for study consent, active upper respiratory infection, airway abnormalities, nasal mass or nasal injury, bleeding disorders, allergies to anesthetics, uncontrolled hypertension, morbid obesity, hepatic or renal failure, cardiovascular diseases, a history of nasopharyngeal surgery and those who were difficult to intubate.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | From Begining of Anesthesia induction to 5th minutes of intubation
Heart rate | From Begining of Anesthesia induction to 5th minutes of intubation
Adverse events | within the first 24 hour after surgery

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT02993692/Prot_SAP_000.pdf